CLINICAL TRIAL: NCT03933319
Title: Phase Ⅱ Study of Pegylated Liposomal Doxorubicin（PLD）Plus Trastuzumab in HER-2 Positive Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Peng Yuan, Principal Investigator, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DMS-BC-11
Record Dates: First submitted 2019-04-29; First posted 2019-05-01 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — liposomal doxorubicin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PLD in combination with trastuzumab (Experimental): Trastuzumab: administered at a loading dose of 8 mg/kg IV followed by 6 mg/kg once every 21 days.
  pegylated liposomal doxorubicin(PLD):administered at dose of 35mg/m2 IV once every 21 days.
  Interventions: Drug: pegylated liposomal doxorubicin

INTERVENTIONS:
Drug: pegylated liposomal doxorubicin — Eligible patients will be treated with the PLD+trastuzumab regimen until the disease progresses or intolerable toxicity

SUMMARY:
This is a single-center phase Ⅱ study designed to evaluated the efficacy and safety of pegylated liposomal doxorubicin（PLD）in combination with trastuzumab in HER-2 positive metastatic breast cancer .

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and voluntarily receive the research procedures according to protocol,willingness to sign the written informed consent document;
* Female patients aged from 18 to 70 years old；
* Histologically confirmed as invasive breast cancer；
* HER-2 Positive（defined by: IHC 3+ or ISH positive）, regardless of HR status;
* Recurrence after adjuvant therapy or metastatic breast cancer，and chemotherapy naïve in the metastatic setting or had one prior regimen for metastatic breast cancer；
* Patients must have measurable disease according to RECIST criteria Version 1.1（Brain metastases lesions and bone metastases lesions were excluded）;
* The adverse event caused by prior therapy has recovered, or stabilized, or does not affect the study administration according to the investigator's judgment；
* Performance status 0-1；
* Life expectancy of at least 3 months；
* Left ventricular ejection fraction (LVEF)≥55%；
* Brain natriuretic peptide (BNP) and cardiac troponin T (cTnT) were in the normal range；
* Patients must have normal ECG；
* Bone marrow function: absolute neutrophil count (ANC)≥1.5×109/L，platelets≥100×109/L，hemoglobin ≥90g/L；
* Hepatic function：alanine aminotransferase(ALT) and aspartate aminotransferase(AST) ≤2.5×ULN，serum total bilirubin≤ 1.5×ULN，or ≤2.5×ULN who has Gilbert's syndrome;
* Renal function：serum creatinine≤1.5×ULN；
* Coagulation function：the international standardized ratio (INR) ≤1.5×ULN, prothrombin time (PT) or the activated partial thrombin time (APTT) ≤1.5×ULN.

Exclusion Criteria:

* Patients with symptomatic brain metastases.
* Patients who are known or suspected to be allergic to the active ingredient or excipients of the investigational drug.
* Prior cumulative dose of 240 mg/m2 for doxorubicin and 400 mg/m2 for epirubicin.
* Prior treatment with anthracyclines has caused cardiotoxicity, or failed (disease progression during therapy or recurrence and metastasis within 12 months after adjuvant therapy).
* Prior mediastinal radiotherapy.
* Participation in other clinical trials within 4 weeks before enrollment.
* Severe cardiovascular disease, including history of congestive heart failure, acute myocardial infarction within 6 months before enrollment, transmural myocardial infarction measured by ECG, uncontrolled arrhythmia, angina requiring therapy, clinically significant valvular heart disease, uncontrolled hypertension.
* Severe or uncontrolled infection.
* Positivity for HIV, Hepatitis B or C.
* Active malignancy in the past 5 years (other than carcinoma in situ of the cervix or basal cell carcinoma of the skin).
* Patients who are pregnant , breastfeeding ,or refuse to use adequate contraception during the course of participation.
* Need to concurrent other cancer therapy(other than palliative care for non-target lesions).
* Other ineligible conditions according to the researcher's judgment.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-03-11 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | approximately 6 months
  The ORR will be calculated as the proportion of patients in the Efficacy Evaluable Patient Set who achieve complete response (CR) and partial response (PR)

SECONDARY OUTCOMES:
Progression-free survival (PFS) | approximately 1.5 years
  PFS will be defined as the time from first dose of study drug until documentation of disease progression or death from any cause
Incidence and Severity of adverse events | approximately 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: peng yuan, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Peng Yuan, Beijing, Beijing Municipality, China